CLINICAL TRIAL: NCT05698654
Title: Evaluation of Longevity Diet and Fasting Mimicking Diet Programs on Body Composition, Disease Risk Factors, and Aging Markers: a Randomized Clinical Trial
Brief Title: Fasting-mimicking Diet and Longevity Diet, Body Composition and Aging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Valter Longo (Other)
Collaborators: University of Calabria (Other); University of Palermo (Other); Regione Calabria / Comune Varapodio (Unknown); IFOM ETS - The AIRC Institute of Molecular Oncology (Other); European Longevity Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-UCALPRG-0004259
Record Dates: First submitted 2023-01-06; First posted 2023-01-26 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-01

CONDITIONS: Overweight; Risk Behavior; Obesity
Keywords: Fasting; Fasting-mimicking diet; Longevity Diet; Longevity; Diet; Aging; FMD; Nutrition; Diseases; LD; Clinical Trial; Randomized; Health; Fat Mass
MeSH Terms: conditions — Overweight; Risk-Taking; Obesity; Fasting; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fasting-mimicking diet (FMD) (Experimental): The fasting-mimicking diet (FMD) group, will be instructed on the benefits and use of the fasting-mimicking diet and how it should be used. This group will have to perform the fasting-mimicking diet once every 3 months (3 cycles in 6 months).
  Interventions: Behavioral: Fasting-mimicking diet (FMD)
- Longevity diet and Fasting-mimicking diet (LD + FMD) (Experimental): This group will undergo both nutritional interventions (LD + FMD); the nutritionist will provide information on the longevity diet andpotential the fasting-mimicking diet, highlighting the advantages of following them. The subjects will be instructed to follow 3 FMD cycles (one cycle every 3 months as for arm 1) combined with the longevity diet plan. The longevity diet includes parts unrelated to diet and involving physical exercise.
  Interventions: Behavioral: Longevity Diet (LD) + Fasting-mimicking Diet (FMD)
- Control Group (No Intervention): Participants in this arm will undergo the same testing as the intervention groups but will be instructed to continue their usual diet. Participants belonging to the control arm will be given an opportunity to follow a 6-month additional LD program starting at the end of 6 months. This trial makes use of a control group to provide robust evidence on the effects of nutritional interventions on the primary and secondary endpoints.

INTERVENTIONS:
Behavioral: Fasting-mimicking diet (FMD) — The subjects will be instructed to follow their usual diet plan, except for 5 days when they eat the foods in the FMD box.The fasting-mimicking diet consists of a blend of 100% plant based nutrients generally regarded as safe. The formulation of these products is based on studies carried out at the Longevity Institute of the University of Southern California and his collaborators over several decades of studies.
  This food plan provides for the replacement of the normal diet with the organic plant products contained in the fasting-mimicking diet for five consecutive days.
  Arms: Fasting-mimicking diet (FMD)
Behavioral: Longevity Diet (LD) + Fasting-mimicking Diet (FMD) — The subjects will be instructed to follow their longevity diet plan, except for 5 days when they eat the foods in the FMD box, based on the following guidelines:
  vegan based diet with the addition of low mercuryfish 2-3 times a week; protein content should be 0.7-0.8 grams per kilogram of ideal weight per day (most of the protein coming from whole cereals,vegetables, legumes and tree nuts only part from fish); monounsaturated and polyunsaturated fats are predominant and very low amounts of saturated and trans-fats are allowed; complex Carbohydrates from vegetables, whole grains and legumes; addition of vitamins, minerals and Omega3 fats; food selected between the traditional food consumed by ancestry; time-restricted feeding: all food must be consumed within 12 hours each day. for those who are overweight or are nearly overweight (BMI >25 kg/m2), either lunch or dinner will be substituted with a low calorie, low sugar snack (approximately 100 kcal: salad, nuts, fruit, etc.).
  Arms: Longevity diet and Fasting-mimicking diet (LD + FMD)

SUMMARY:
This study was designed as a large, randomized, controlled clinical trial in a heterogeneous population and is aimed at assessing as a primary objective whether the fasting-mimicking diet alone or in combination with the longevity diet can modify the percentage of fat mass in a cohort of subjects stratified by sex, age and body mass index. As secondary objectives, will evaluate the effects of the fasting-mimicking diet alone or in combination with the longevity diet on the general health conditions of the population.

From a public health point of view, the efficacy of a food intervention such as the longevity diet and/or short periods of fasting-mimicking diet would represent proof of the results that can be achieved by a realistics, feasible and inexpensive approach.

The information obtained is relevant because the nutritional intervention will be undertaken by people who live in their normal environment and who simply receive every day dietary guidelines, and support and/or boxes containing a 5 day meal program to be consumed in lieu of their normal diet once every 3 months.

DETAILED DESCRIPTION:
This is a randomized, open-label in adult subjects: arm 1 will include subjects randomized to follow a Fasting Mimicking Diet (FMD) plan with a 5-day meal program once every two months for a 6-month period (3 cycles); arm 2 will include subjects randomized to follow the FMD plus a Longevity Diet (LD) program for a 6-month period (FMD+LD); arm 3 will include randomized to the control group that will be recommended to continue their usual diet. Participants belonging to the control arm will be given an opportunity to follow a 6-month LD program starting at the end of 6 months.

Recruitment

Participants with BMI >=25 kg/m2 and in the 30 to 65 year range will be identified in towns within of a range of 20 km from Varapodio (province of Reggio Calabria, Southern Italy).The confirmation of eligibility and subsequent consenting will be carried out at the screening visit.

Eligible participants will undergo 5 different visits (pre-screening visit, screening visit, baseline visit (t0), and two follow-up visits (after 3 and 6 months from the baseline visit). Participants belonging to the control arm who decide to follow an optional 6-month LD program at the last follow-up visit (month 6), will receive two additional visits at month 9 and at month 12.

Pre-screening phone call visit

The purpose of the pre-screening visit is to determine if a potential participant fits the study's core inclusion criteria (age and BMI) and doesn't meet some of its permanent exclusion criteria (e.g. morbidities, pregnancy, known allergies, etc.). Once a potential participant is cleared through the pre-screening visit and confirms interest in participating, he/she may proceed to the screening visit.

Screening visit

The purpose of the screening visit is to confirm the volunteer's eligibility for study participation. Participants who meet all inclusion/exclusion criteria, will be informed about the research study before any procedure is performed. Participants must provide written informed consent to the processing of personal data in an anonymous and aggregate form in compliance with the requirements of the EU General Data Protection Regulation 2016/679 (GDPR) and the relevant Italian laws implementing the GDPR, including the Legislative Decree No.101/2018 of 10 August 2018 on the protection of privacy in relation to the processing of personal data. Any collection, processing and disclosure of personal data, such as participant health and medical information is subject to compliance with the aforementioned personal data protection laws.

Screening will include measurement of height, weight, and vital signs, review of medical history and current medications, assessment of sleep quality and disturbances and collection of fasting blood. Participants will be then randomized into either one of the intervention arms (FMD or FMD+LD) or in the control arm using a web-based randomization system that will be controlled by the researchers of the Valter Longo Foundation in Milan

Baseline visit (T0)

Within a week from the screening visit, subjects in arm 1 and 2 (FMD or FMD+LD) will be given the box of FMD together with ketone test strips to self-monitor urinary ketone bodies during the FMD cycles. Subjects in arm 2 will be given informative material and instructions for the LD. During the visit, staff will administer the questionnaire for assessing life style and dietary habits. The baseline visit will also include body composition assessment using Bioelectrical Impedance Analysis (BIA), measurement of height, weight, and vital signs, medical history, current medications and a collection of fasting blood. Blood testing information will be also retried from the screening visit.

A portion of subjects for each study group reporting a sleep problem on the basis of the score obtained at the Pittsburgh Sleep Quality Index (PSQI) questionnaire will also receive an Oura Ring device for the continuous monitoring of sleep state and wakefulness. These three study groups will be balanced for age, sex, BMI and for the score obtained at the PSQI.

Visit 2 (after three months or 5-7 days after the second FMD cycle, T1)

After 3 months from the randomization, subjects in the FMD and FMD+LD arms will be contacted to receive the FMD boxes for the second and the third FMD cycles, respectively, together with the ketone test strips to self-monitor urinary ketone bodies during the FMD cycles. Visit 2 will also include body composition assessment using BIA, measurement of height, weight, and vital signs and to assess sleep quality and disturbances.

Visit 3 (after six months or 5-7 days after the third FMD cycle,T2)

During the clinical visit, staff will assess signs and symptoms of adverse events, review compliance to the diet programs. Visit 3 will also include body composition assessment using BIA, measurement of height, weight, and vital signs, medical history and current medications and a collection of fasting blood for both hematological and genetic analyses as previously described for the baseline visit. Only subjects who undergo home sleep monitoring at the baseline visit will also receive an Oura Ring device for the continuous monitoring of sleep state and wakefulness. After this period, study staff will assess sleep quality and disturbances with the PSQI and will answer any questions from the subject. At this point, subjects belonging to the control arm will be given an opportunity to follow a LD program for a 6-month period (optional).

Optional visit at month 9 and 12

Subjects belonging to the arm 3 who decide to follow an optional LD program for a 6-month period after the end of the study at 6 months will meet with the study nutritionist during the clinical visits at month 9 and month 12. Staff will review compliance to the LD program and answer any questions by the subject.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of 30-65 years of age;
* Body mass index equal to or greater than 25 kg/m2.

And at least one of the following:

* Obesity (Body mass index equal to or greater than 30 kg/m2).
* HbA1C greater than 5.6%;
* IGF-1 level greater than 200 ngml-1;
* Systolic blood pressure >130 mmHg and diastolic blood pressure >90 mmHg;
* Triglycerides >150 mgdl-1;
* C-reactive protein >1 mgL-1;
* Total cholesterol >190 mgdL-1 and LDL cholesterol >129 mgdL-1.

Exclusion Criteria:

* individuals with a family member already included in the study;
* individuals who are allergic to tree nuts (macadamia, cashew, almond, pecan), soy, oats, sesame, or celery/celeriac;
* pregnant females;
* Individuals with any documented cancer diagnosis within the past 5 years;
* documented myocardial infarction within past 5 years;
* documented cerebrovascular accident within past 5 years;
* chronic steroid use (longer than 45 consecutive days);
* insulin-dependent diabetes mellitus;
* individuals taking insulin or insulin-like drugs and individuals taking hypoglycemic agents other than metformin. In this last case, close attention will therefore be paid to the self-monitoring of blood glucose during the FMD cycles;
* Individuals with severe hypertension (systolic greater than 200 mmHg and or diastolic greater than 105 mmHg.

  * Change in prescription medications, over-the-counter (OTC) medications, medical foods, and nutritional supplements within 30 days prior to the start and for the duration of the study.
  * Use of medications classified as narcotics 15 days prior start and for the duration of the study.
  * Use of prescription medications and/or over-the-counter medications for acute and semi- acute medical conditions 15 days prior to start and for the duration of the study.
  * Use of acetaminophen is permitted on an as-needed basis.
  * Use of an investigational drug or participation in an investigational study within 30 days prior to the start and for the duration of the study.
  * Use of oral or injectable corticosteroids within 30 days prior to the start and for the duration of the study.
  * Use of anticoagulant medications (heparin compounds or warfarin) within 30 days prior to the start and for the duration of the study. Use of aspirin 81 mg or 325 mg once daily is permitted.
  * Use of neuroactive prescription medications including major and atypical antipsychotic medications, anti-depressants, anti-anxiolytics, and epilepsy medications within 30 days prior to the start and for the duration of the study.

(subjects will not be allowed to discontinue prohibited prescription medications to meet enrolment criteria).

* A history of allergy or intolerance to study products. Detailed descriptions of study product are included in Section 4.1 and 4.2, appended to the Study Informed Consent.
* Clinically significant vital sign abnormalities (systolic blood pressure <90 mmHg or >200 mmHg, diastolic blood pressure <50 mmHg or >105 mmHg or resting heart rate of <50 or >100 bpm) at screening visit.
* A serious, unstable illness including cardiac, hepatic, renal, gastrointestinal, respiratory, endocrinologic, neurologic, immunologic, or hematologic disease.
* Known infection with HIV, TB or Hepatitis B or C.
* A current diagnosis or personal history of:

  * Any cardiovascular disease including myocardial infarction, angina, cardiovascular surgery (within 5 years), congestive heart failure, cardiac arrhythmias or conduction abnormalities, cerebrovascular accident, transient ischemic attack (TIA), or peripheral vascular disease, deep vein thrombosis or pulmonary embolus. Diabetes mellitus requiring inhaled or injected insulin.
  * Any autoimmune disease such as inflammatory bowel disease (including Crohn's disease and/or ulcerative colitis), multiple sclerosis, rheumatoid arthritis, systemic lupus erythematosus, polymyositis, scleroderma and/or thyroiditis.
  * Any significant liver or kidney disease such as cirrhosis or non-alcoholic fatty liver disease, glomerulonephritis, and/or ongoing dialysis treatment.
  * Any malignancy (with the exception of adequately treated malignancies with no known recurrence for >2 years).
* Any serious mental illness including a history of attempted suicide.
* Any medical condition that in the opinion of the primary care doctor or a specialist would preclude safe participation in this study or interfere with compliance.
* Use of drugs of abuse (such as marijuana, cocaine, phencyclidine [PCP] and methamphetamine) 15 days prior to Day 1 and for the duration of the study.
* History of regular intake of >14 alcoholic drinks per week for females, and >21 drinks per week for males (1 drink = 35 cl. beer, 12 cl. wine, or 30 ml. hard liquor).

Technical reasons

Any condition in which bioelectrical impedance testing would be impossible or uninterpretable (e.g. prostheses in extremities on both sides, limb amputation, implanted pacemaker, inability to lay still or supine, or skin defects on preferred electrode placement sites.

Other Exclusion Criteria: Inability to comply with study and/or follow-up visits.

* Any concurrent condition (including clinically significant abnormalities in medical history, physical examination or laboratory evaluations) which, in the opinion of the PI, would preclude safe participation in this study or interfere with compliance.
* Any sound medical, psychiatric and/or social reason which, in the opinion of the PI, would preclude safe participation in this study or interfere with compliance.
* Abnormal laboratory findings including: abnormal blood counts (hematocrit < 33% or > 47%; WBC < 3.0 or > 12.0 x10^3/mm3; platelets < 140 or > 500 x 10^9/L); abnormal kidney function test (creatinine > 2.5 mg/dL) or liver function test(s) (AST, ALT, alkaline phosphatase) > 1.5X the upper limit of normal; serum calcium > 11 mg/dL); serum K < 3.5 mEq/L; Na < 134 or > 148 mmolL-1

Women of Childbearing Potential Contraception: the effects of the study products on the developing human fetus have not been studied extensively. For this reason, women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Females of childbearing potential will have a pregnancy test prior to receiving study products. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform study staff and her primary care physician immediately.

Pregnancy: because there is an unknown but potential risk for adverse events in pregnant women during treatment with the study products, pregnant women are not eligible for study participation.

Breast-feeding: Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study products, breastfeeding mothers are not eligible for study participation.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 501 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Body Fat Percentage | Comparison of the clinical marker up to 7 days after the randomization and 6 months after the randomization (6 months)
  Change from baseline to end of study in body composition measured as percentage of fat mass.

SECONDARY OUTCOMES:
Change of blood glucose values | Comparison of the clinical marker up to 7 days after the randomization and 6 months after the randomization (6 months)
  (mg / dl)
Change of blood insulinemic values | Comparison of the clinical marker up to 7 days after the randomization and 6 months after the randomization (6 months)
  (µU/mL)
Change of blood glycated hemoglobin | Comparison of the clinical marker up to 7 days after the randomization and 6 months after the randomization (6 months)
  (percentage)
Change of blood LDL, HDL, total cholesterol and triglycerides | Comparison of the clinical marker up to 7 days after the randomization and 6 months after the randomization (6 months)
  (mg/dl)
Change of blood pressure | Comparison of the clinical marker up to 7 days after the randomization and 6 months after the randomization (6 months)
  (mmHg)
Change of body weight | Comparison of the clinical marker up to 7 days after the randomization and 6 months after the randomization (6 months)
  (Kg)
Change of BMI | Comparison of the clinical marker up to 7 days after the randomization and 6 months after the randomization (6 months)
  (kg/m^2)
Change of telomere length | Comparison of the clinical marker up to 7 days after the randomization and 6 months after the randomization (6 months)
  (kb)
Change in Pittsburgh Sleep Quality Index | Comparison of the clinical marker up to 7 days after the randomization and 6 months after the randomization (6 months)
  (PSQI)
Change in Berlin questionnaire | Comparison of the clinical marker up to 7 days after the randomization and 6 months after the randomization (6 months)
  (Berlin questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Romina Inès Cervigni, Study Director — Fondazione Valter Longo; Alberto Montesanto, Study Chair — Department of Biology, Ecology and Earth Sciences, University of Calabria
Locations (1):
- Ambulatorio Medico presso Biblioteca Comunale, Varapodio, Calabria, Italy

REFERENCES:
- [Background] Knoops KT, de Groot LC, Kromhout D, Perrin AE, Moreiras-Varela O, Menotti A, van Staveren WA. Mediterranean diet, lifestyle factors, and 10-year mortality in elderly European men and women: the HALE project. JAMA. 2004 Sep 22;292(12):1433-9. doi: 10.1001/jama.292.12.1433. PMID 15383513
- [Background] Brandhorst S, Choi IY, Wei M, Cheng CW, Sedrakyan S, Navarrete G, Dubeau L, Yap LP, Park R, Vinciguerra M, Di Biase S, Mirzaei H, Mirisola MG, Childress P, Ji L, Groshen S, Penna F, Odetti P, Perin L, Conti PS, Ikeno Y, Kennedy BK, Cohen P, Morgan TE, Dorff TB, Longo VD. A Periodic Diet that Mimics Fasting Promotes Multi-System Regeneration, Enhanced Cognitive Performance, and Healthspan. Cell Metab. 2015 Jul 7;22(1):86-99. doi: 10.1016/j.cmet.2015.05.012. Epub 2015 Jun 18. PMID 26094889
- [Background] Houston M, Hays L. Acute effects of an oral nitric oxide supplement on blood pressure, endothelial function, and vascular compliance in hypertensive patients. J Clin Hypertens (Greenwich). 2014 Jul;16(7):524-9. doi: 10.1111/jch.12352. Epub 2014 Jun 24. PMID 24962851
- [Background] Gallus S, Odone A, Lugo A, Bosetti C, Colombo P, Zuccaro P, La Vecchia C. Overweight and obesity prevalence and determinants in Italy: an update to 2010. Eur J Nutr. 2013 Mar;52(2):677-85. doi: 10.1007/s00394-012-0372-y. Epub 2012 May 27. PMID 22645105
- [Background] Wei M, Brandhorst S, Shelehchi M, Mirzaei H, Cheng CW, Budniak J, Groshen S, Mack WJ, Guen E, Di Biase S, Cohen P, Morgan TE, Dorff T, Hong K, Michalsen A, Laviano A, Longo VD. Fasting-mimicking diet and markers/risk factors for aging, diabetes, cancer, and cardiovascular disease. Sci Transl Med. 2017 Feb 15;9(377):eaai8700. doi: 10.1126/scitranslmed.aai8700. PMID 28202779
- [Background] Levine ME, Suarez JA, Brandhorst S, Balasubramanian P, Cheng CW, Madia F, Fontana L, Mirisola MG, Guevara-Aguirre J, Wan J, Passarino G, Kennedy BK, Wei M, Cohen P, Crimmins EM, Longo VD. Low protein intake is associated with a major reduction in IGF-1, cancer, and overall mortality in the 65 and younger but not older population. Cell Metab. 2014 Mar 4;19(3):407-17. doi: 10.1016/j.cmet.2014.02.006. PMID 24606898
- [Background] Pollack MN. Insulin, insulin-like growth factors, insulin resistance, and neoplasia. Am J Clin Nutr. 2007 Sep;86(3):s820-2. doi: 10.1093/ajcn/86.3.820S. PMID 18265475

DOCUMENTS (2):
  • Study Protocol (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT05698654/Prot_000.pdf
  • Informed Consent Form (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT05698654/ICF_001.pdf